CLINICAL TRIAL: NCT06849024
Title: Effect of Transcutaneous Electrical Nerve Stimulation on Proinflammatory Cytokines, Angiogenic and Growth Factors in Subjects with Venous Ulcers of the Lower Extremities: a Clinical Trial
Brief Title: Electrostimulation in Patients with Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario de Tonalá (Other)
Collaborators: Diabetes sin complicaciones S.A de C.V (Unknown); Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Arieh Roldán Mercado Sesma, Associate B professor, Centro Universitario de Tonalá
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TENS-EC01-2021
Record Dates: First submitted 2025-02-13; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2023-04

CONDITIONS: Venous Leg Ulcer
Keywords: leg venous ulcers; TENS; electrical stimulation
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A Electrostimulation (Experimental): Transcutaneous electrical nerve stimulation or placebo during 30 minutes three times per week for 60 days.
  Interventions: Device: Transcutaneous electrical neurostimulation
- Group B Placebo (Sham Comparator): Transcutaneous electrical nerve stimulation without stimulation during 30 minutes three times per week for 60 days.
  Interventions: Device: Transcutaneous electrical neurostimulation

INTERVENTIONS:
Device: Transcutaneous electrical neurostimulation — Transcutaneous electrical nerve stimulation or placebo during 30 minutes three times per week for 60 days.

SUMMARY:
Abstract Evaluate the effect of transcutaneous electrical nerve stimulation on proinflammatory cytokines, angiogenic and growth factors in subjects with venous ulcers of the lower extremities.

Material and Methods A randomized, double-blind, placebo-controlled, parallel-groups clinical trial was carried out in 32 adults (18-75 years of age) with venous ulcers of the lower extremities according to CEAP classification with duple Doppler ultrasound. After random allocation of intervention 16 patients received continuous and intermittent transcutaneous electrical nerve stimulation or placebo during 30 minutes three times per week for 60 days. Proinflammatory cytokines, angiogenic and growth factors were measured before and after intervention. Mann-Whitney U test and Wilcoxon's rank-sum test were performed to statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Venous ulcers C6,Es, As/Ap,Pr according to CEAP classification by Spanish Society of Angiology and Vascular Surgery or demonstrated with duplex Doppler ultrasound
* Who did not respond to conventional treatment.
* Evolution of no less than 12 weeks
* Ulcers with a size > 2 and < 12 cm in any of its dimensions did not affect the dermis and epidermis, but should not spread to the tendon or bone, without formation of ischemia and infection.

Exclusion Criteria:

* Patients with active superficial or deep thrombus phlebitis, chronic arterial insufficiency (figures less than 0.8 in IPTB), neoplasms.
* Treated with chemotherapy or radiation therapy
* Clinically infected ulcers at the time of study evaluation, signs of cellulitis.
* Osteomyelitis or ulcer with a necrotic background Individuals with a surgical history of venous insufficiency at least 12 months prior to undergoing the protocol.
* Participants with diseases such as rheumatoid arthritis, lupus erythematosus, or disseminated, mental diseases, electrical implants (bypass), pregnancy and breastfeeding, diabetes mellitus, lung cancer, a history of stroke, or undergoing anticoagulant treatment.
* Patients receiving corticosteroids or some other immunosuppressive, non-steroidal anti-inflammatory, histamine antagonists, or antibiotics on a regular basis within 4 weeks prior to the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Changed in plasma concentration from baseline of pro-inflammatory cytokines, angiogenic and growth factors in subjects with venous ulcers of the lower extremities | From the beginning of treatment at 60 days
  Changed in plasma concentration from baseline of EGF, VEGF, PDGF-BB, TNF-, IL-1, IL-6, TSP-1 and TIMP-1 and 2 from basa to 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Medico Nacional de Occidente. Hospital de Especialidades. Instituto Mexicano del Seguro Social, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No